CLINICAL TRIAL: NCT00079001
Title: A Randomized Double-Blind, Placebo-Controlled Phase III Study of Early Versus Standard Zoledronic Acid to Prevent Skeletal Related Events in Men With Prostate Cancer Metastatic to Bone
Brief Title: Zoledronate in Preventing Skeletal (Bone)-Related Events in Men Who Are Receiving Androgen Deprivation Therapy For Prostate Cancer and Bone Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Eastern Cooperative Oncology Group (Network); NCIC Clinical Trials Group (Network); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CALGB-90202; U10CA031946 (NIH); CAN-NCIC-PRC2; CDR0000353209 (Registry Identifier: NCI Physician Data Query); NCT00698308 (obsolete NCT alias)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer; bone metastases
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Zoledronic Acid; Androgen Antagonists; Gonadotropin-Releasing Hormone; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronic acid + androgen deprivation therapy (Experimental): 4mg by IV over 15 minutes every 4 weeks in the absence of disease progression or the first skeletal-related event. Participants who progression on blinded treatment before having a skeletal event may continue on open label Zoledronic acid (4 mg by IV over 15 minutes every 3 weeks).
  Interventions: Drug: zoledronic acid; Drug: androgen deprivation therapy; Drug: GnRH agonist; Dietary Supplement: Calcium supplement; Dietary Supplement: Vitamin D
- Placebo + androgen deprivation therapy (Active Comparator): Placebo bu IV over 15 minutes for 4 weeks in the absence of disease progression or the first skeletal-related event. Participants who progress on blinded treatment before having a skeletal event may continue on open label Zoledronic acid.
  Interventions: Other: placebo; Drug: androgen deprivation therapy; Drug: GnRH agonist; Dietary Supplement: Calcium supplement; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: zoledronic acid — Given IV
  Arms: Zoledronic acid + androgen deprivation therapy
Other: placebo — Given IV
  Arms: Placebo + androgen deprivation therapy
Drug: androgen deprivation therapy — Patients concurrently enrolled on the Phase III study of intermittent androgen deprivation in patients with stage D2 prostate cancer will receive androgen deprivation therapy per SWOG-9346. All other patients will receive androgen deprivation therapy at a standard dose and schedule throughout the study.
Drug: GnRH agonist — Patients concurrently enrolled on the Phase III study of intermittent androgen deprivation in patients with stage D2 prostate cancer will receive the GnRH agonist per SWOG-9346. All other patients will receive GnRH agonist at a standard dose and schedule throughout the study.
Dietary Supplement: Calcium supplement — Patients will receive 500 mg by mouth daily of a calcium supplement or a combination tablet containing approximately 500 mg elemental calcium and 400-500 IU vitamin D by mouth daily.
Dietary Supplement: Vitamin D — Patients will receive a multivitamin tablet containing 400-500 IU vitamin D by mouth daily or a combination tablet containing approximately 500 mg elemental calcium and 400-500 IU vitamin D by mouth daily.

SUMMARY:
RATIONALE: Zoledronate may prevent or decrease skeletal (bone)-related events (such as pain or fractures) caused by bone metastases and androgen deprivation therapy. It is not yet known whether treatment with zoledronate is effective in preventing bone-related events in patients who have prostate cancer and bone metastases.

PURPOSE: This randomized phase III trial is studying how well zoledronate works in preventing bone-related events in patients who are receiving androgen deprivation therapy for prostate cancer and bone metastases.

DETAILED DESCRIPTION:
Zoledronic acid decreases the risk of skeletal related events in men with prostate cancer metastatic to bone and disease progression after primary hormonal therapy.

This study is designed to evaluate whether earlier treatment with zoledronic acid will further decrease the risk of skeletal related events. This is a randomized, double-blind, placebo-controlled, multicenter study followed by an open-label study. Patients are stratified according to ECOG performance status (0-1 vs 2), prior skeletal-related event (no vs yes), and serum alkaline phosphatase (< upper limit of normal [ULN] vs ≥ ULN).

The primary objective of the study is to determine whether treatment with zoledronic acid at the time of initiation of androgen deprivation therapy for metastatic prostate cancer will delay the time to first skeletal related event. The secondary objective of the study is to compare the effect of treatment with zoledronic acid to placebo on overall survival (OS), progression-free survival (PFS) and toxicity in men receiving androgen deprivation therapy for metastatic prostate cancer.

Patients are randomized to 1 of 2 treatment arms. Treatment continues in the absence of disease progression or a skeletal-related event. All patients receive concurrent androgen deprivation therapy with a GnRH agonist. Patients also receive oral calcium and (vitamin D) supplements daily. Patients progressing to androgen-independent prostate cancer proceed to the open-label therapy with zoledronic acid IV. Treatment continues for 3 weeks in the absence of disease progression or the first skeletal-related event.

Patients are followed periodically for approximately 10 years after entry on the study.

ELIGIBILITY:
1. Histologic Documentation: Histologic documentation of prostate adenocarcinoma. Patients with small cell, neuroendocrine, or transitional cell carcinomas are not eligible.
2. Staging: At least one bone metastasis by radiographic imaging (bone scan, magnetic resonance imaging, computed tomography, or plain radiographs). Indeterminate lesions should be confirmed by a second imaging method. Imaging to document bone metastases is to be completed either within 12 weeks before registration or within 12 weeks before initiating androgen deprivation therapy for bone metastases.
3. Hormone Therapy

   * While on this study, patients must receive androgen deprivation therapy (ADT) for treatment of prostate cancer. Androgen deprivation therapy may have begun prior to enrollment on this study; however patients must have initiated ADT ≤ 6 months prior to enrollment.
   * Androgen deprivation therapy is defined as bilateral orchiectomy or gonadotropin- releasing hormone (GnRH) agonist with or without an antiandrogen.
   * Patients treated with intermittent androgen deprivation therapy are not eligible except for patients concurrently enrolled in SWOG-9346/INT-0162/CALGB 9594, Phase III Study of Intermittent Androgen Deprivation in Patients with Stage D2 Prostate Cancer.
4. Prior Treatment:

   * Hormone therapy at any point prior to 6 months before enrollment is prohibited. This includes any of the following treatments:

     * orchiectomy,
     * GnRH agonist (e. g., leuprolide, goserelin, triptorelin),
     * estrogen therapy,
     * antiandrogen (e. g., bicalutamide, flutamide, nilutamide), or
     * any other therapy known to lower testosterone level or inhibit testosterone effect.
   * Prior neoadjuvant and/or adjuvant hormone therapy is allowed provided that the duration of hormone therapy was six months or less and the hormone therapy was discontinued more than 6 months prior to study entry.
   * No prior treatment with a bisphosphonate
   * No prior treatment with denosumab
   * No prior treatment with radiopharmaceuticals
   * ≥ 4 weeks since completion of prior radiation therapy with at least one bone metastasis present that has NOT been radiated.
5. ECOG (CTC) performance status 0-2
6. Age: ≥ 18 years
7. Required Initial Laboratory Data:

   * Calculated Creatinine Clearance ≥ 30 mL/min
   * Corrected serum calcium ≥ 8.0 mg/dL (2.00 mmol/L) and <11.6 mg/dL (2.90 mmol/L)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2004-01; Primary Completion 2012-07 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R. Smith, MD, PhD, Study Chair — Massachusetts General Hospital
Locations (241):
- United States (238):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Loma Linda (Pettis), Loma Linda, California
  - Pismo Beach, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Ruby L. Golleher Cancer Program at Presbyterian Intercommunity Hospital, Whittier, California
  - Yale Cancer Center, New Haven, Connecticut
  - Veterans Affairs Medical Center - West Haven, West Haven, Connecticut
  - Kaiser Permanente at Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Leesburg Regional Medical Center, Leesburg, Florida
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Heartland Oncology and Hematology, Council Bluffs, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Iowa City, Iowa City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Union Memorial Hospital, Baltimore, Maryland
  - Good Samaritan Hospital of Maryland, Baltimore, Maryland
  - Kaiser Permanente at Woodlawn Medical Center, Baltimore, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - John R. Marsh Cancer Center at Washington County Hospital, Hagerstown, Maryland
  - Kaiser Permanente Mid-Atlantic Medical Group-Largo Medical Facility, Largo, Maryland
  - Kaiser Permanente Capital Area Medical Group - Shady Grove Facility, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - Duke Health Raleigh Hospital, Raleigh, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Wood County Oncology Center, Bowling Green, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Susquehanna Cancer Center at Divine Providence Hospital, Williamsport, Pennsylvania
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Self Regional Cancer Center at Self Regional Medical Center, Greenwood, South Carolina
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - St. Luke's Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Kaiser Permanente Medical Center - Fair Oaks, Fairfax, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Wheaton Franciscan Cancer Care - St. Joseph, Milwaukee, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (3):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario

REFERENCES:
- [Result] Smith MR, Halabi S, Ryan CJ, Hussain A, Vogelzang N, Stadler W, Hauke RJ, Monk JP, Saylor P, Bhoopalam N, Saad F, Sanford B, Kelly WK, Morris M, Small EJ. Randomized controlled trial of early zoledronic acid in men with castration-sensitive prostate cancer and bone metastases: results of CALGB 90202 (alliance). J Clin Oncol. 2014 Apr 10;32(11):1143-50. doi: 10.1200/JCO.2013.51.6500. Epub 2014 Mar 3. PMID 24590644
- [Derived] Jakob T, Tesfamariam YM, Macherey S, Kuhr K, Adams A, Monsef I, Heidenreich A, Skoetz N. Bisphosphonates or RANK-ligand-inhibitors for men with prostate cancer and bone metastases: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 3;12(12):CD013020. doi: 10.1002/14651858.CD013020.pub2. PMID 33270906
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2004 and May 2012, 645 participants were registered and randomized.
Period: Overall Study
Arm/Group | Zoledronic Acid + Androgen Deprivation Therapy | Placebo + Androgen Deprivation Therapy
Started | 323 | 322
Completed | 323 | 322
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid + Androgen Deprivation Therapy | Placebo + Androgen Deprivation Therapy | Total
Number analyzed (Participants) | 323 | 322 | 645
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.1 [60.0 to 72.5] | 66.7 [60.2 to 73.6] | 66.3 [60.0 to 73.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 323 | 322 | 645
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 42 | 50 | 92
  White | 261 | 256 | 517
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 323 | 321 | 644
  Canada | 0 | 1 | 1
ECOG Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  participants
    0 | 205 | 205 | 410
    1 | 105 | 105 | 210
    2 | 13 | 12 | 25
Prior Skeletal Related Event [Number; unit: participants]
  Yes | 42 | 40 | 82
  No | 281 | 282 | 563

OUTCOME MEASURES:

1. Primary Outcome: Time to First Skeletal Related Event
Description: Time to first skeletal related event (SRE) was defined as the time from randomization to first skeletal event. Skeletal events are defined as radiation to bone, clinical fracture, surgery to bone and spinal cord compression and death due to prostate cancer. The median with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Up to 10 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zoledronic Acid + Androgen Deprivation Therapy | Placebo + Androgen Deprivation Therapy
Number analyzed (Participants) | 323 | 322
months | 31.9 [24.2 to 40.3] | 28.8 [25.3 to 37.2]
Statistical Analysis 1: Comparison: Zoledronic Acid + Androgen Deprivation Therapy vs Placebo + Androgen Deprivation Therapy; The null hypothesis was that the hazard ratio is greater than or equal to 1.0 versus the alternative hypothesis that the hazard ratio is less than 0.77. With a target of 470 SREs, log-rank statistic had 88% power to detect a 23% decrease in hazard of SRE (equivalent to an increase in median time to SRE from 30 months to 39 months), assuming a one-sided type I error rate of .05; Test type: Non-Inferiority or Equivalence — Superiority and futility analysis were conducted for time to first SRE. Lan-Demets analog of the Emerson-Fleming sequential boundary was used to maintain overall significance level of α = .05 while conducting interim analyses on time to first SRE; p = 0.385, Log Rank — Because of early termination, conditional power was performed under the alternative hypothesis. This is the probability that zoledronic acid is superior to placebo, given time to first SRE data at interim analysis under alternative hypothesis; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0 to 1.174] — Patients randomly assigned to zoledronic acid were compared with patients assigned to placebo

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from randomization to death of any cause. Surviving patients were censored at the date of last follow-up. The median OS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Up to 10 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zoledronic Acid + Androgen Deprivation Therapy | Placebo + Androgen Deprivation Therapy
Number analyzed (Participants) | 323 | 322
months | 37.9 [34.2 to 49.2] | 36.0 [30.2 to 41.6]
Statistical Analysis 1: Comparison: Zoledronic Acid + Androgen Deprivation Therapy vs Placebo + Androgen Deprivation Therapy; Test type: Superiority or Other; p = 0.29, Log Rank; Adjusted for stratification factors: performance status, prior SRE, and serum alkaline phosphatase; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.70 to 1.12] — Zoledronic acid versus placebo group

3. Secondary Outcome: Progression-free Survival
Description: Progression Free Survival (PFS) was defined as the time from registration until disease progression or death, whichever occurs first. The median PFS with 95% CI was estimated using the Kaplan-Meier method.
  Progression is defined as one or more of the following: new bone metastases, biochemical progression of PSA, treatment with radiation therapy while on treatment.
Time Frame: Up to 10 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zoledronic Acid + Androgen Deprivation Therapy | Placebo + Androgen Deprivation Therapy
Number analyzed (Participants) | 323 | 322
months | 10.6 [8.5 to 15.4] | 9.2 [8.0 to 11.9]
Statistical Analysis 1: Comparison: Zoledronic Acid + Androgen Deprivation Therapy vs Placebo + Androgen Deprivation Therapy; Test type: Superiority or Other; p = 0.22, Log Rank; Adjusted for stratification factors: performance status, prior SRE, and serum alkaline phosphatase; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.74 to 1.07] — Zoledronic acid versus placebo group

ADVERSE EVENTS:
Description: All patients that reported adverse events were used to summarize the adverse events, data is available on 618 participants. Participants that were not assessed for adverse events were not included in the adverse event table.
Arm/Group | Zoledronic Acid + Androgen Deprivation Therapy | Placebo + Androgen Deprivation Therapy
Serious Adverse Events (participants affected / at risk) | 60/310 | 61/308
Other Adverse Events (participants affected / at risk) | 269/310 | 266/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid + Androgen Deprivation Therapy (N=310) | Placebo + Androgen Deprivation Therapy (N=308)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (9) | 6 (6)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac disorder (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac pain (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 2 (5)
Myocardial ischemia (Cardiac disorders) | 5 (5) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Endocrine disorder (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 10 (10) | 7 (7)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (14) | 18 (21)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (10) | 14 (16)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 5 (5) | 2 (2)
Death NOS (General disorders) | 1 (1) | 1 (1)
Disease progression (General disorders) | 3 (3) | 3 (3)
Edema limbs (General disorders) | 1 (3) | 3 (4)
Fatigue (General disorders) | 33 (39) | 32 (42)
Fever (General disorders) | 5 (5) | 5 (5)
General symptom (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 3 (3) | 2 (2)
Sudden death (General disorders) | 3 (3) | 1 (1)
Bladder infection (Infections and infestations) | 2 (3) | 2 (3)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Urethral infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (4)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0)
Coagulopathy (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 22 (25) | 18 (19)
INR increased (Investigations) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 2 (2) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (2) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 2 (2)
Weight loss (Investigations) | 0 (0) | 2 (3)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 16 (18) | 18 (21)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 18 (21) | 18 (21)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 6 (7)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 10 (11) | 8 (8)
Serum potassium decreased (Metabolism and nutrition disorders) | 16 (16) | 9 (10)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (18) | 22 (27)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Oculomotor nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 3 (5) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 2 (2)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Kidney pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 5 (5) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 3 (4) | 0 (0)
Ureteric perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 7 (7) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Thrombosis (Vascular disorders) | 1 (1) | 4 (4)
Vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid + Androgen Deprivation Therapy (N=310) | Placebo + Androgen Deprivation Therapy (N=308)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (14) | 6 (6)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 1 (1)
Edema (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (7) | 0 (0)
Cataract (Eye disorders) | 3 (3) | 2 (3)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (10)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 61 (148) | 52 (127)
Diarrhea patients with a colostomy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 70 (150) | 78 (209)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Salivary gland disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 40 (59) | 41 (67)
Chest pain (General disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 37 (64) | 25 (55)
Disease progression (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 191 (1076) | 193 (1232)
Fever (General disorders) | 43 (56) | 29 (42)
Gait abnormal (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (4) | 1 (1)
Hypersensitivity (Immune system disorders) | 8 (12) | 6 (22)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Infection without neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 3 (3) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 1 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Venous injury - Extremity-upper (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (3)
Alkaline phosphatase increased (Investigations) | 16 (25) | 13 (21)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 77 (299) | 65 (316)
Laboratory test abnormal (Investigations) | 3 (6) | 1 (1)
Leukocyte count decreased (Investigations) | 6 (6) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 2 (8) | 2 (5)
Neutrophil count decreased (Investigations) | 4 (4) | 3 (4)
Platelet count decreased (Investigations) | 1 (2) | 2 (4)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 2 (5)
Anorexia (Metabolism and nutrition disorders) | 54 (128) | 58 (128)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 13 (23) | 11 (25)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 3 (7)
Serum calcium decreased (Metabolism and nutrition disorders) | 59 (109) | 56 (113)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 23 (34) | 28 (100)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 38 (101) | 38 (79)
Serum potassium decreased (Metabolism and nutrition disorders) | 44 (108) | 36 (89)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 6 (7) | 5 (5)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (12) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (32) | 8 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 20 (32) | 21 (30)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (8) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (11)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 166 (849) | 140 (680)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (6) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 8 (11) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (6) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 1 (1)
Mini mental status examination abnormal (Nervous system disorders) | 1 (17) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (2)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (13) | 3 (3)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Kidney pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Kidney perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (4) | 5 (12)
Urinary retention (Renal and urinary disorders) | 3 (6) | 4 (7)
Urogenital disorder (Renal and urinary disorders) | 1 (4) | 2 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 10 (42) | 5 (46)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (3) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (20)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (12)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (70) | 25 (79)
Rash desquamating (Skin and subcutaneous tissue disorders) | 36 (74) | 47 (120)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 4 (11) | 3 (5)
Hypertension (Vascular disorders) | 4 (8) | 5 (11)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.